CLINICAL TRIAL: NCT00329329
Title: Phase 1 Study of the Oral Platinum Agent Satraplatin in Combination With Capecitabine for the Treatment of Patients With Advanced Solid Malignancies
Brief Title: Study of Satraplatin With Capecitabine to Treat Advanced Solid Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decided to discontinue study drug development
Sponsor: Agennix (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAT1-05-02
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Malignancies
Keywords: Advanced solid malignancies
MeSH Terms: conditions — Neoplasms | interventions — satraplatin; Capecitabine

INTERVENTIONS:
Drug: satraplatin and capecitabine — satraplatin and capecitabine dose escalated per the dosing scheme

SUMMARY:
The purpose of this study is to determine the maximally tolerated dose (MTD) and Phase 2 recommended dose of satraplatin when administered in combination with capecitabine in patients with advanced solid malignancies.

DETAILED DESCRIPTION:
This is a single center, open-label, non-randomized, Phase I dose finding study of the investigational, oral cytotoxic drug, satraplatin in combination with capecitabine in patients with advanced solid tumors for whom curative therapy is not available. Please refer to the Eligibility Criteria below for key inclusion and exclusion criteria.

PURPOSE: The purpose of this trial is to determine a tolerable dose and schedule for the combination of satraplatin and docetaxel when given to patients with advanced solid tumors.

WHAT IS SATRAPLATIN: Satraplatin is an oral, investigational anticancer drug that is a member of the platinum-based class of chemotherapy drugs. Platinum-based drugs have been clinically proven to be one of the most effective classes of anticancer therapies. Unlike the currently marketed platinum-based drugs, satraplatin can be given orally.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed solid tumor that is metastatic or unresectable and for which standard curative or palliative chemotherapy measures do not exist or are no longer effective
* Age > 18 years old
* ECOG Performance Status < 2
* Female patients may not be pregnant or lactating and must be willing to practice contraception
* Adequate organ function as defined by the following:

  * Serum creatinine < 1.5 mg/dl
  * Absolute neutrophil count (ANC) > 1500/dL
  * Platelets > 100,000/dL
  * Total bilirubin < upper limit of normal (ULN) for the reference lab
  * AST, ALT, and alkaline phosphatase must be within the designated range allowing for eligibility

Key Exclusion Criteria:

* Other chemotherapy treatment < 4 weeks prior to enrollment Treatment with capecitabine, 5-fluorouracil (5-FU), or a platinum agent < 3 months from time of enrollment
* Radiotherapy involving > 30% of the active bone marrow
* Radiotherapy < 4 weeks prior to enrollment
* Pre-existing peripheral neuropathy > grade 1
* Pre-existing hearing loss > grade 2
* Metastatic brain or meningeal tumors unless the patient is > 6 months from definitive therapy, had a negative imaging study within 4 weeks of study entry, is clinically stable with respect to the tumor at the time of study entry, and is not receiving steroid therapy or taper
* Patients who have not recovered (> grade 1) from the following toxicities of previous regimens before enrollment:

  * hematologic toxicities
  * fatigue
  * mucositis
  * nausea/vomiting
  * diarrhea
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)
* Uncontrolled intercurrent illness including, but not limited to, ongoing active infection, uncontrolled congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness that would limit compliance with study requirements
* History of hypersensitivity reaction to capecitabine, 5-FU or any platinum containing drugs
* History of human immunodeficiency (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
* Evidence of concurrent second malignancy other than basal cell carcinoma of the skin or cervical carcinoma in situ
* Concurrent use of medications that inhibit cytochrome P450 3A4 (including aprepitant)
* History of bone marrow or major organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-05; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
MTD | 2007

SECONDARY OUTCOMES:
Safety | 2007

CONTACTS AND LOCATIONS:
Overall Officials: William Gradishar, MD, Principal Investigator — Northwestern University Medical Center
Locations (1):
- Northwestern University Medical Center, Chicago, Illinois, United States